CLINICAL TRIAL: NCT01949324
Title: A Phase 2 Multicenter Randomized Clinical Trial of Ciliary Neurotrophic Factor (CNTF) for Macular Telangiectasia Type 2 (MacTel)
Brief Title: A Phase 2 Multicenter Randomized Clinical Trial of CNTF for MacTel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Collaborators: The Lowy Medical Research Institute Limited (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTMT-02
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Macular Telangiectasia Type 2
Keywords: MacTel
MeSH Terms: interventions — Ciliary Neurotrophic Factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- NT-501 Implant procedure (Experimental): The investigational product is the NT-501 encapsulated cell system which consists of cells encapsulated within a semi-permeable polymer membrane and supportive matrices. NT-501 contains NTC-201 cells that were derived from the NTC-200 cell line by genetic modification so as to secrete recombinant human ciliary neurotrophic factor (CNTF).
  Interventions: Biological: Ciliary neurotrophic factor (CNTF); Device: NT-501 Implant; Procedure: NT-501 Implant procedure
- Sham procedure (Sham Comparator): Non-penetrating sham procedure to mimic implant procedure
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Biological: Ciliary neurotrophic factor (CNTF) — Ciliary neurotrophic factor released from NT-501 encapsulated cell implant
  Arms: NT-501 Implant procedure
Procedure: Sham procedure — Sham surgery for Sham arm
  Arms: Sham procedure
Device: NT-501 Implant — NT-501 encapsulated cell implant
  Arms: NT-501 Implant procedure
Procedure: NT-501 Implant procedure — Surgery to implant device for NT-501 encapsulated cell implant releasing human ciliary neurotrophic factor arm
  Arms: NT-501 Implant procedure

SUMMARY:
This study is a phase 2, randomized, multi-center, single-masked study to evaluate the efficacy and safety of the NT-501 implants in participants with Mactel.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be offered sufficient opportunity to review and to understand the informed consent form, agree to the form's contents and sign the protocol's informed consent
* Participant must have at least one study eye with a positive diagnosis of MacTel Type 2
* Participant must have an IS/OS PR break in the study eye(s) and en face ellipsoid zone (area of IS/OS loss) as measured by SDOCT between 0.16 mm2 and 4.00 mm2
* If female, participant must be incapable of pregnancy
* If male, participant must agree to use an effective form of birth control during the study

Exclusion Criteria:

* Participant is unable to provide informed consent
* Participant is less than 21 years of age or greater than 80 years of age
* Participant is medically unable to comply with study procedures or follow-up visits
* Participant was a study subject in any other clinical trial of an intervention (drug or device) within the last 6 months
* Participant is pregnant or breastfeeding

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-04; Primary Completion 2017-04-14 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Ellipsoid zone (area of IS/OS loss) as measured by en face imagining by SDOCT in study eye(s) | 24 months
  Change in the ellipsoid zone (area of IS/OS loss) from baseline to month 24 as measured by en face imaging by SDOCT in study eye(s)

SECONDARY OUTCOMES:
Ellipsoid zone | 12 months
  Change in the ellipsoid zone from baseline to Month 12.
Retinal sensitivity (dB) as measured by microperimetry | 12 and 24 months
  Change in retinal sensitivity (dB) as measured by microperimetry from baseline to Months 12 and 24.
Increase in ellipsoid zone | 12 and 24 months
  Proportion of study eyes with a 35% or more increase from baseline in the ellipsoid zone at Months 12 and 24.
Visual Acuity | 12 and 24 months
  Change in best corrected visual acuity (BCVA) from baseline to Months 12 and 24.
Visual Acuity | 12 and 24 Months
  Proportion of study eyes with 15 or more letter loss from baseline in BCVA at Months 12 and 24.
Visual Acuity | 12 and 24 Months
  Proportion of study eyes with 10 or more letter loss from baseline in BCVA at Months 12 and 24.
Reading Speed | 12 and 24 Months
  Change in reading speed as measured by the IReST from baseline to Months 12 and 24.

OTHER OUTCOMES:
Cone density as measured by AOSLO | 12 and 24 Months
  Change in cone density as measured by AOSLO from baseline to Months 12 and 24, in selected participants.
National Eye Institute Visual Functioning Questionnaire | 12 and 24 months
  Change in NEI VFQ (overall and subscale) from baseline to Months 12 and 24.
Electroretinogram changes | 6, 12 and 24 Months
  Electroretinogram (ERG) changes from baseline to Months 6, 12 and 24, in selected clinics/participants.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - Jules Stein Eye Institute, Los Angeles, California
  - Bascom Palmer, Miami, Florida
  - Emory University, Atlanta, Georgia
  - National Eye Institute, Bethesda, Maryland
  - Massachusetts Eye and Ear Infirmary, Retina Service, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - University of Wisconsin, Madison, Wisconsin
- Australia (3):
  - Save Sight Institute, Sydney, New South Wales
  - Centre for Eye Research Australia, East Melbourne
  - Lions Eye Institute, Nedlands

REFERENCES:
- [Derived] Loo J, Cai CX, Choong J, Chew EY, Friedlander M, Jaffe GJ, Farsiu S. Deep learning-based classification and segmentation of retinal cavitations on optical coherence tomography images of macular telangiectasia type 2. Br J Ophthalmol. 2022 Mar;106(3):396-402. doi: 10.1136/bjophthalmol-2020-317131. Epub 2020 Nov 23. PMID 33229343